CLINICAL TRIAL: NCT02617628
Title: Improving Outcomes of Opioid Addicted Prisoners With Extended-Release Injectable Naltrexone (Vivitrol) Before vs. After Reentry
Brief Title: Outcomes of Opioid Addicted Prisoners With Extended-Release Injectable Naltrexone
Acronym: OAPXRNTX
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FC14-1409-21688
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Opiate Dependence
Keywords: opioid addiction
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Before Re-entry (Active Comparator): Extended Release Naltrexone, 380 mg injection, 1x monthly for 4 months
  Interventions: Drug: extended release naltrexone
- After Re-entry (Active Comparator): Extended Release Naltrexone, 380 mg injection, 1x monthly for 4 months
  Interventions: Drug: extended release naltrexone

INTERVENTIONS:
Drug: extended release naltrexone — Extended Release Naltrexone is currently marketed in the US for use in adults with alcohol dependence. It will be administered in this study at the currently marketed dose of 380 mgs. Subjects will be randomized to receive one injection of 380 mg of extended release naltrexone, at baseline, before they leave the prison, or either 380 mg of extended release naltrexone after they are released from prison. Both groups will receive three additional monthly doses of 380 mgs while enrolled in intensive outpatient treatment for six months. Subjects will also receive weekly psychosocial counseling.
  Other Names: Vivitrol

SUMMARY:
This study is a collaboration between the University of Pennsylvania, the Philadelphia Prison System, and the North East Treatment Center (NETSteps). It purpose is to study the impact of an injectable opiate addiction medication (extended release naltrexone) given before reentry into the community that might help to improve reconnection to healthcare and other support systems, and possibly help reduce recidivism.

DETAILED DESCRIPTION:
The primary objectives for this study is to offer tools to support improve healthcare and related outcomes and reduce the risk of relapse and recidivism for opiate addicted prisoners reentering into the community after release from correctional facilities. In this study the investigators examine a medication-assisted therapy (extended release naltrexone) that is likely to be acceptable to correctional facilities and opioid addicted prisoners and that can improve the outcomes achieved by the usual detoxification/treatment referral approach. The results may be used to facilitate policy changes that involve adding extended release naltrexone to correctional facility formularies for use before reentry, and collaborating with one or more outpatient treatment providers to maintain continuity of care. Two hundred (200) opioid addicted prisoners currently incarcerated in the Philadelphia Prison System, who meet study admission criteria and express an interest in extended release naltrexone treatment, who give informed consent and will be scheduled for release within 14 days of being randomized into the study will be enrolled. These 200 subjects will be stratified by sex (male/females), will be 18 years or older, and are not sentenced).

ELIGIBILITY:
Inclusion Criteria:

* Opioid dependent with physiological features according to Diagnostic and Statistical Manual of Mental Disorders-5th edition
* Interested in extended release naltrexone treatment
* Eligible to have health benefits reinstated
* Detoxified and able to pass a naloxone challenge (e.g. no withdrawal within 30 minutes after receiving 0.8 mg naloxone I.M. and documented by a score <5 on the Clinical Opiate Withdrawal Scale
* Age 18 or above
* Not being transferred to serve a longer sentence in a State or Federal prison
* Provide their address or phone number along with the names and contact information of 3 or more persons likely to know where they can be reached with permission to contact them if unable to be reached in other ways
* Able to speak and read English and provide informed consent
* able to correctly answer 9 of 10 study quiz items
* not pregnant and agree to the use of an acceptable form of birth control
* can access to NET Steps via car or public or other transportation after reentry

Exclusion Criteria:

* Planning to move from the Philadelphia area within the next 6 months
* Neurological, cardiovascular, renal, hepatic (Alanine aminotransferase, Aspartate aminotransferase or Gamma-glutamyl transpeptidase >3 times top limit of normal) or another medical disorder that seriously impairs or makes hazardous ability to participate
* Active tuberculosis
* Currently psychotic, homicidal, suicidal
* Uncontrolled seizure disorder
* History of allergy to naltrexone, polylactide-co-glycolide, carboxymethylcellulose, or any other components of the diluent
* Chronic pain for which opioids are needed
* Sentenced to naltrexone Treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George E Woody, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center on the Studies of Addiction, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Cadet T, Jalali A, Jeng PJ, Poole S, Woody G, Murphy SM. Determinants of health-related quality of life among individuals with opioid use disorder, recently released from incarceration. Addict Sci Clin Pract. 2023 May 25;18(1):34. doi: 10.1186/s13722-023-00375-0. PMID 37231479

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started August 2016 and ended June 16, 2018 in the Philadelphia Prison System. Subjects all were recruited while incarcerated.
Pre-assignment Details: Subjects were stratified to sentenced/not sentenced and male/female
Groups:
- Before Re-entry: Extended Release Naltrexone, 380 mg injection
  Subjects will be randomized to receive one injection of 380 mg of extended release naltrexone, at baseline (month 1), before they leave the prison. Subjects will also receive one injection 380 mg of extended-release naltrexone at month 2, month 3, and month 4. Subjects will receive weekly psychosocial counseling for six months.
- After Re-entry: Extended Release Naltrexone, 380 mg injection
  Subjects will be randomized to receive one injection of 380 mg of extended release naltrexone, at baseline (month 1), after they leave the prison. Subjects will also receive one injection 380 mg of extended-release naltrexone at month 2, month 3, and month 4. Subjects will receive weekly psychosocial counseling for six months.
Period: Overall Study
Arm/Group | Before Re-entry | After Re-entry
Started | 74 | 72
Completed | 12 | 11
Not Completed | 62 | 61
Not completed — Withdr, Transfers-other prisons, dropout | 62 | 61

BASELINE CHARACTERISTICS:
Groups:
- After Re-entry: Extended Release Naltrexone, 380 mg injection, 1x monthly for 4 months
  Extended release naltrexone: Extended Release Naltrexone is currently marketed in the US for use in adults with alcohol dependence. It was administered in this study at the currently marketed dose of 380 mgs. Subjects were randomized to receive one injection of 380 mg of extended release naltrexone after they were released from prison. Both groups received three additional monthly doses of 380 mgs while enrolled in intensive outpatient treatment for six months. Subjects also received weekly psychosocial counseling.
- Before Re-entry: Extended Release Naltrexone, 380 mg injection, 1x monthly for 4 months
  Extended release naltrexone: Extended Release Naltrexone is currently marketed in the US for use in adults with alcohol dependence. It was administered in this study at the currently marketed dose of 380 mgs. Subjects were randomized to receive one injection of 380 mg of extended release naltrexone, at baseline, before they left the prison. Both groups received three additional monthly doses of 380 mgs while enrolled in intensive outpatient treatment for six months. Subjects also received weekly psychosocial counseling.
- Total: Total of all reporting groups
Arm/Group | After Re-entry | Before Re-entry | Total
Number analyzed (Participants) | 74 | 72 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 72 | 146
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (10.0) | 36.2 (8.5) | 37.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 54 | 52 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 18 | 37
  Not Hispanic or Latino | 55 | 54 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 10 | 29
  White | 54 | 61 | 115
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 74 | 72 | 146
Opioid Drug Use [Count of Participants; unit: Participants] — The number of subjects who used opioids, including heroin, in the past 30 days at baseline
  Participants | 74 | 72 | 146
EuroQol Overall Health [Count of Participants; unit: Participants] — Mobility measures walking ability. score =0 to 3, with 0= no problem, 1=slight problems, and 2=moderate problems, and 3=severe problems. X=Did not want to answer.
  Participants
    Mobility: No Problems | 69 | 60 | 129
    Mobility: Slight Problems | 3 | 4 | 7
    Mobility: Moderate Problems | 1 | 7 | 8
    Mobility: Severe Problems | 1 | 0 | 1
    Mobility: x=Missing | 0 | 1 | 1
    Self Care: No Problems | 71 | 67 | 138
    Self Care: Slight Problems | 2 | 2 | 4
    Self Care: Moderate Problems | 1 | 2 | 3
    Self Care: Severe Problems | 0 | 0 | 0
    Self Care: x=Missing | 0 | 1 | 1
    Doing Usual Activities: No Problems | 65 | 59 | 124
    Doing Usual Activities: Slight Problems | 5 | 8 | 13
    Doing Usual Activities: Moderate Problems | 4 | 3 | 7
    Doing Usual Activities: Severe Problems | 0 | 1 | 1
    Doing Usual Activities: x=Missing | 0 | 1 | 1
    Pain or Discomfort: No Problems | 42 | 35 | 77
    Pain or Discomfort: Slight Problems | 15 | 20 | 35
    Pain or Discomfort: Moderate Problems | 13 | 12 | 25
    Pain or Discomfort: Severe Problems | 4 | 4 | 8
    Pain or Discomfort: x=Missing | 0 | 1 | 1
    Anxiety and Depression: No Problems | 18 | 21 | 39
    Anxiety and Depression: Slight Problems | 27 | 22 | 49
    Anxiety and Depression: Moderate Problems | 15 | 21 | 36
    Anxiety and Depression: Severe Problems | 14 | 7 | 21
    Anxiety and Depression: x=Missing | 0 | 1 | 1
Beck Depression Index [Count of Participants; unit: Participants]
  No Depression | 44 | 39 | 83
  Clinical Depression | 30 | 31 | 61
  Missing | 0 | 2 | 2
Timeline Follow-Back [Mean (Standard Deviation); unit: days] — Mean Days of drug use past 30 days before baseline
  days
    Heroin Use | 21.91 (12.6) | 25.56 (9.59) | 23.71 (11.3)
    Methadone Use | .92 (4.7) | 1.19 (4.9) | 1.05 (4.7)
    Other Opioids | 8.46 (12.05) | 6.97 (11.06) | 7.73 (11.56)
    Benzodiazepines | 6.36 (10.59) | 7.78 (11.11) | 7.06 (10.84)
    Cocaine | 12.7 (13.01) | 14.19 (13.27) | 13.44 (13.11)
Risk Assessment Battery [Mean (Standard Deviation); unit: units on a scale] — Seventeen items make-up scores for Drug-Risk and Sex-Risk in the Risk Assessment Battery (RAB). Drug-Risk is scored from 0 to 22. Sex-Risk is scored from 0 to18. Total Score = Total Drug Risk + Total Sex-Risk. The overall "Total Score" is then divided by 40, the highest possible score. Items are not differentially weighted. Higher values reflect greater frequency of risky behavior.
  units on a scale
    Drug Risk Score | 3.19 (4.33) | 4.42 (4.87) | 3.79 (4.6)
    Sex Risk Scoe | 5.61 (2.89) | 5.94 (2.66) | 5.77 (2.77)
    Total RAB Score | 8.80 (6.17) | 10.36 (6.68) | 9.57 (6.45)

OUTCOME MEASURES:

1. Primary Outcome: Relapse to Opioid Use in Subjects by Month 3
Description: Proportion (count) without relapse by month 3 post release. At each monthly assessment we determined whether a subject relapsed based on the timeline follow-back (TLFB) and/or urine drug screen results (UDS) and self-reported withdrawal.
Time Frame: 12 weeks (month 3)
Population: In treatment arm 1 (before reentry) 38 subjects received vivitrol before leaving prison.
  In treatment arm 2 (after reentry) 48 subjects were eligible to receive injections after release from prison. Arm 2 subjects were to return to the research clinic within 7 days after release to receive their first injection.
Measure: Count of Participants; unit: Participants
Groups:
- Before Re-entry: Extended Release Naltrexone, 380 mg injection
  Subjects will be randomized to receive one injection of 380 mg of extended release naltrexone, at baseline (month 1), before they leave the prison. Subjects will also receive one injection 380 mg of extended-release naltrexone at month 2, month 3, and month 4. Subjects will receive weekly psychosocial counseling for six months.
  intensive outpatient treatment for six months. Subjects also received weekly psychosocial counseling.
- After Re-entry: Extended Release Naltrexone, 380 mg injection
  Subjects will be randomized to receive one injection of 380 mg of extended release naltrexone, at baseline (month 1), After they leave the prison. Subjects will also receive one injection 380 mg of extended-release naltrexone at month 2, month 3, and month 4. Subjects will receive weekly psychosocial counseling for six months.
  outpatient treatment for six months. Subjects also received weekly psychosocial counseling.
Arm/Group | Before Re-entry | After Re-entry
Number analyzed (Participants) | 38 | 48
Participants | 16 | 20
Statistical Analysis 1: Comparison: Before Re-entry vs After Re-entry; Based on Lee et al. we estimated a 23-33% group difference in relapse by month 3. Power estimates calculated this estimate with a 2-sided alpha of .05 and a baseline sample size of 100 per group resulted in 80% power to detect a difference of approximately 20% (OR = 2.4) between groups assuming a rate of 50% in the control condition and 10% and 20% attrition by 3- and 6-month follow-ups. For the 86 participants randomized and released, with 80% power; and odds ratio of 3.5; Test type: Equivalence — The odds ratio for relapse versus non-relapse for the AR group relative to the BR group was analyzed, as well as the corresponding odds ratio for unknown relative to non-relapse; p = 0.38, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.57 to 4.27] — Threshold for significance was set at p<.05

2. Secondary Outcome: Reincarceration
Description: percentage of patients who were reincarcerated
Time Frame: 0 to 28 months
Population: This outcome was determined as follows: one XR-NTX injection provided 4 weeks of treatment. Study patients also had counseling, thus weeks in treatment equaled the weeks of protected time from XR-NTX plus the number of weeks a patient had one or more counseling appointments after the protection from the last XR-NTX dose ended.
Measure: Count of Participants; unit: Participants
Arm/Group | Before Re-entry | After Re-entry
Number analyzed (Participants) | 38 | 48
Participants | 28 | 22
Statistical Analysis 1: Comparison: Before Re-entry vs After Re-entry; We used Cox proportional hazards regression model to compare the groups on time to reincarceration; Test type: Superiority; p = 0.01, Regression, Cox; Cox Proportional Hazard = -0.74486

ADVERSE EVENTS:
Time Frame: 2 years, 2 months
Description: The definition is the same as clinicaltrials.gov.
  Collection:
  Medical staff evaluated the intensity, seriousness, and causal relationship of the AE to study medication and procedures. The research medical staff asked the participant what adverse events have occurred since the last visit. Medical Staff evaluated for relatedness to study interventions. If serious, IRBs were notified in 5 days and followed up to determine its outcome.
Groups:
- Before Re-entry: Extended Release Naltrexone, 380 mg injection, 1x monthly for 4 months
  Extended Release Naltrexone is currently marketed in the US for use in adults with alcohol dependence. It will be administered in this study at the currently marketed dose of 380 mgs. Subjects will be randomized to receive one injection of 380 mg of extended release naltrexone, at baseline, before they leave the prison. Both groups will receive three additional monthly doses of 380 mgs while enrolled in intensive outpatient treatment for six months. Subjects will also receive weekly psychosocial counseling.
- After Re-entry: Extended Release Naltrexone, 380 mg injection, 1x monthly for 4 months
  Extended Release Naltrexone is currently marketed in the US for use in adults with alcohol dependence. It will be administered in this study at the currently marketed dose of 380 mgs. Subjects will be randomized to receive one injection of 380 mg of extended release naltrexone after they are released from prison. Both groups will receive three additional monthly doses of 380 mgs while enrolled in intensive outpatient treatment for six months. Subjects will also receive weekly psychosocial counseling.
Arm/Group | Before Re-entry | After Re-entry
All-Cause Mortality (participants affected / at risk) | 1/74 | 3/72
Serious Adverse Events (participants affected / at risk) | 10/74 | 13/72
Other Adverse Events (participants affected / at risk) | 35/74 | 21/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Before Re-entry (N=74) | After Re-entry (N=72)
overdose (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (9)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
kidney pain (Renal and urinary disorders) | 2 (2) | 0 (0) — kidney stone
panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
broken rib (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Before Re-entry (N=74) | After Re-entry (N=72)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 6 (6) | 3 (3)
anxiousness (Psychiatric disorders) | 5 (5) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
back pain-lower (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
nose bleed (General disorders) | 0 (0) | 1 (1)
blurry vision (Eye disorders) | 1 (1) | 0 (0)
achey joints (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
allergy in left eye (Eye disorders) | 0 (0) | 1 (1)
arthritis in leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
body aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
chest pain-cardiac (Cardiac disorders) | 1 (1) | 1 (1)
common cold (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
depression (Psychiatric disorders) | 5 (7) | 2 (2)
injection site reaction (General disorders) | 8 (12) | 4 (5)
malaise (Immune system disorders) | 2 (2) | 4 (4)
diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
headache (Nervous system disorders) | 6 (6) | 3 (3)
toothache (Gastrointestinal disorders) | 6 (8) | 1 (1)
breathing problems (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 2 (2)
wrist pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
nausea with vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
flu like symptoms (Immune system disorders) | 0 (0) | 2 (2)
eye infection (Infections and infestations) | 0 (0) | 1 (1)
suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
decreased sex drive (Reproductive system and breast disorders) | 0 (0) | 1 (1)
fibrois mass on ovary (Reproductive system and breast disorders) | 1 (1) | 0 (0)
increased urine (Renal and urinary disorders) | 1 (1) | 0 (0)
hip and left femor ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
infected boil (Infections and infestations) | 1 (1) | 0 (0)
heart burn (Gastrointestinal disorders) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
insect bite swelling (Immune system disorders) | 1 (1) | 0 (0)
accidental inury, arm and knuckle (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
excessive sweating (General disorders) | 1 (1) | 0 (0)
withdrawn feeling (Psychiatric disorders) | 1 (1) | 0 (0)
foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
hernia pain (General disorders) | 0 (0) | 1 (1)
hip arthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
hot-cold sweats (General disorders) | 1 (1) | 0 (0)
irritable (Psychiatric disorders) | 1 (1) | 0 (0)
lethargic (General disorders) | 0 (0) | 1 (1)
miscarriage of pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
muscle ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (3)
restless (Nervous system disorders) | 0 (0) | 1 (1)
runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
breathing abnormality (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
sore throat (Gastrointestinal disorders) | 1 (1) | 0 (0)
tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT02617628/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT02617628/ICF_001.pdf